CLINICAL TRIAL: NCT00202137
Title: A Randomized Controlled Trial of the Effects of Home Blood Pressure Monitoring on Blood Pressure Control
Brief Title: Home Blood Pressure Monitoring and Blood Pressure Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Principal Investigator, Dr. Richard Birtwhistle, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBPM; HSFO Grant # T-5345 (Other Grant/Funding Number: Ontario Heart and Stroke Foundation)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
Keywords: Home Blood Pressure, Hypertension, Blood Pressure Control
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): home blood pressure monitoring with automatic blood pressure device
  Interventions: Behavioral: Home blood pressure monitoring
- 2 (Active Comparator): physician monitoring of blood pressure by 3 monthly office visits
  Interventions: Behavioral: Physician monitoring of blood pressure

INTERVENTIONS:
Behavioral: Home blood pressure monitoring — Monitor blood pressure using home blood pressure monitor
  Arms: 1
Behavioral: Physician monitoring of blood pressure — Blood pressure measured as standard care from physician (no home monitor given for blood pressure monitoring)
  Arms: 2

SUMMARY:
Hypertension is a common problem in Canada with a prevalence of about 15%. The goal of hypertension therapy should be to maximize blood pressure control. Home blood pressure monitoring (HBPM) devices are available and many patients are using them. The role that self-monitoring of blood pressure can play in optimizing blood pressure control is unclear. We hope to clarify the role of home blood pressure monitoring in the treatment of hypertension and explore how it may affect patient and physician behaviours related to blood pressure management. This study will compare a group of hypertensive patients who use HBPM with those who do not use these devices. The intervention (HBPM) group will measure their blood pressure at home a minimum of once weekly and will report these measurements to their family doctor at each visit. The control group will receive usual care as delivered by their family doctor. Outcomes of blood pressure control will be measured over a 12 month period. Outcomes will be determined primarily by 24 hour ambulatory blood pressure monitoring and by reviewing data in patient's charts located in family physicians office. Fifty family physicians from the Kingston area have agreed to participate.

DETAILED DESCRIPTION:
The objective of this study is to measure the effect of home (self) blood pressure monitoring on control of hypertension in a primary care setting.

This research is important for several reasons:

i) Lack of control of hypertension is common and is associated with morbidity and mortality.

ii) The costs of managing hypertensions are high, not only because of the prevalence of hypertension, but also because maintenance of control must exist over many years for most patients.

iii) Home blood pressure monitoring is increasingly being used by patients.

iv) Guidelines for home blood pressure monitoring are already being developed and distributed.

v) While it would seem helpful to increase self-care by patients, there is currently conflicting or inadequate evidence that home monitoring is useful.

The main hypothesis of the study is that, compared to patients who receive usual care, patients who use home monitoring will have lower blood pressure levels.

Our secondary hypothesis is that HBPM changes physician and patient behaviours in ways that would result in better control of hypertension.

The methodology uses cluster randomization. Physicians will be randomly allocated to either have their patients use the intervention or to continue with usual care. The intervention for the experimental group is the provision of a home blood pressure monitor to patients with a request that they record weekly blood pressure measurements and report them to their family physician at their regular hypertension follow-up visits. The physicians will be informed of current guidelines for target levels for home monitored blood pressure. The control group will receive usual care.

The main outcome measures will be blood pressure level (by 24 hour ambulatory monitoring) at baseline, 6 months and 12 months.

The secondary objective of this study is to measure the effect of home monitoring on physicians' and patients' behaviours related to hypertension control. Behaviours that will be measured include the intensity and type of pharmacological treatment, compliance with antihypertensive medication and changes in patient's lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* adults age 18 years and older with essential hypertension.
* who are treated with medication to lower their blood pressure.
* whose mean daytime blood pressure at enrolment is 135/85 mm Hg or greater.
* and who are not currently using HBPM.

Exclusion Criteria:

* a diagnosis of secondary hypertension.
* pregnancy.
* hypertension management primarily by a consultant.
* a disability that precludes use of a home blood pressure monitor.
* enrolled in another hypertension trial
* white coat hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2002-07; Primary Completion 2007-04 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The mean nighttime blood pressures on ABPM. | 6mth and 1yr
Achieving BP target at end of study | 6mt and 1yr

SECONDARY OUTCOMES:
patient lifestyle changes. | 6mth and 1yr
the number of visits for hypertension. | 6mth & 1yr
compliance with hypertensive medication use | 6month & 1yr
compliance with the intervention | 6month & 1yr
intensity of treatment | 6month & 1yr
frequency of lifestyle counseling by physician | 6month & 1yr
Quality of Life as measured by SF-36. | 6month & 1yr

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Godwin, MD MSc, Principal Investigator — Queen's University, Kingston, Ontario, Canada; Richard Birtwhistle, MD MSc, Principal Investigator — Queen's University, Kingston, Ontario, Canada
Locations (1):
- Centre for Studies in Primary Care, Kingston, Ontario, Canada

REFERENCES:
- [Background] Godwin M, Ruhland L, Casson I, MacDonald S, Delva D, Birtwhistle R, Lam M, Seguin R. Pragmatic controlled clinical trials in primary care: the struggle between external and internal validity. BMC Med Res Methodol. 2003 Dec 22;3:28. doi: 10.1186/1471-2288-3-28. PMID 14690550
- [Background] Beckett L, Godwin M. The BpTRU automatic blood pressure monitor compared to 24 hour ambulatory blood pressure monitoring in the assessment of blood pressure in patients with hypertension. BMC Cardiovasc Disord. 2005 Jun 28;5(1):18. doi: 10.1186/1471-2261-5-18. PMID 15985180
- See also: An article describing the methodology — http://www.biomedcentral.com/1471-2288/3/28